CLINICAL TRIAL: NCT03699449
Title: An uMbrella Study of BIomarker-driven Targeted Therapy In Patients With Platinum-resistant Recurrent OvariaN Cancer(AMBITION)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Collaborators: AstraZeneca (Industry); Samsung Genomic Institute (Unknown); Seoul National University Hospital (Other); Samsung Medical Center (Other); Korean Gynecologic Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0749; KCT0003283 (Other: CRIS); KGOG3045 (Other: KGOG); 2018-10-009 (Other: Samsung Medical Center); 1810-035-977 (Other: Seoul National Univ. Hosp); ESR-17-12678 (Other: AstraZeneca)
Record Dates: First submitted 2018-10-02; First posted 2018-10-09 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Platinum-resistant Recurrent Ovarian Cancer
MeSH Terms: interventions — durvalumab; tremelimumab

STUDY DESIGN:
Intervention Model Description: This is a randomized, multi-center, open label, phase II study for HRD+ patients and a biomarker-driven multiple-arm phase II study for HRD- patients.
  This study will consist of a number of study modules (substudies), each evaluating the antitumor activity of targeted agents in patients whose tumors express specific phenotype relevant to the molecules under investigation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- olaparib + cediranib (Experimental): olaparib+cediranib combination therapy
  Interventions: Drug: olaparib+cediranib combination therapy
- durvalumab + olaparib (Experimental): durvalumab + olaparib combination therapy
  Interventions: Drug: durvalumab + olaparib combination therapy
- durvalumab + chemotherapy (Experimental): durvalumab +chemotherapy
  Interventions: Drug: durvalumab + chemotherapy treatment
- durvalumab + tremelimumab + chemotherapy (Experimental): durvalumab + tremelimumab + chemotherapy
  Interventions: Drug: durvalumab + tremelimumab + chemotherapy treatment
- durvalumab + tremelimumab + paclitaxel (Experimental): durvalumab + tremelimumab + paclitaxel
  Interventions: Drug: durvalumab + tremelimumab + paclitaxel treatment
- durvalumab +chemotherapy (Experimental): durvalumab +chemotherapy
  Interventions: Drug: durvalumab +chemotherapy treatment

INTERVENTIONS:
Drug: olaparib+cediranib combination therapy — Cediranib (30mg p.o. qd) + Olaparib (200mg p.o. bid) until disease progression
  Arms: olaparib + cediranib
Drug: durvalumab + olaparib combination therapy — Durvalumab (1500mg i.v. every 4 weeks starting on week 5 day1 for up to 12 months) + Olaparib (300mg p.o. bid) until disease progression
  Arms: durvalumab + olaparib
Drug: durvalumab + chemotherapy treatment — Durvalumab (1500mg i.v. every 4 weeks for up to 24 months) + non-platinum-based standard of care chemotherapy (weekly paclitaxel, topotecan, or Pegylated liposomal doxorubicin(PLD) up to 6 cycles)
  Chemotherapy regimen:
  Weekly Paclitaxel 80mg/m2 (day 1,8,15,22 every 4 weeks), PLD (40mg/m2 on D1 every 4 weeks), topotecan (4mg/m2 on D1,8,15 every 4 weeks)
  Arms: durvalumab + chemotherapy
Drug: durvalumab + tremelimumab + chemotherapy treatment — Durvalumab (1500mg i.v. every 4 weeks for up to 24 months) + Tremelimumab (75mg i.v. every 4 weeks for up to 4 doses) + non-platinum-based standard of care chemotherapy (weekly paclitaxel, topotecan, or Pegylated liposomal doxorubicin (PLD) up to 4 cycles)
  Chemotherapy regimen:
  Weekly Paclitaxel 80mg/m2 (day 1,8,15,22 every 4 weeks), PLD (40mg/m2 on D1 every 4 weeks), topotecan (4mg/m2 on D1,8,15 every 4 weeks)
  Arms: durvalumab + tremelimumab + chemotherapy
Drug: durvalumab + tremelimumab + paclitaxel treatment — Durvalumab (1500mg i.v. every 4 weeks for up to 24 months) + Tremelimumab (300mg i.v. once) + non-platinum-based standard of care chemotherapy (weekly paclitaxel up to 4 cycles)
  Chemotherapy regimen:
  Weekly Paclitaxel 60mg/m2 (day 1,8,15 every 4 weeks)
  Arms: durvalumab + tremelimumab + paclitaxel
Drug: durvalumab +chemotherapy treatment — Durvalumab (1500mg i.v. every 4 weeks for up to 24 months) + non-platinum-based standard of care chemotherapy (paclitaxel, topotecan, or Pegylated liposomal doxorubicin(PLD) up to 4 cycles)
  Chemotherapy regimen:
  Weekly Paclitaxel 80mg/m2 (day 1,8,15,22 every 4 weeks), PLD (40mg/m2 on D1 every 4 weeks), topotecan (4mg/m2 on D1,8,15 every 4 weeks)
  Arms: durvalumab +chemotherapy

SUMMARY:
This study is a pilot study of biomarker-driven targeted therapy in patients with platinum-resistant recurrent ovarian cancer. More specifically, this is a randomized, multi-center, open label, phase II study for Homologous Recombination Deficiency(HRD)+ patients and a biomarker-driven multiple-arm phase II study for Homologous Recombination Deficiency(HRD)- patients.

This study will consist of a number of study modules (substudies), each evaluating the antitumor activity of targeted agents in patients whose tumors express specific phenotype relevant to the molecules under investigation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high-grade serous or high-grade endometrioid ovarian, primary peritoneal, or fallopian tube cancers.
* Disease progression within 6 months of completing platinum-based chemotherapy
* Who had received ≥ two lines of chemotherapy
* Provision of informed consent prior to any study specific procedures
* Female aged 20 years older at time of study entry
* Body weight >30kg
* Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below: 1) Haemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days, 2) Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, 3) Platelet count ≥ 100 x 109/L, 4) Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN), 5) Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 3 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤ 5x ULN, 6) Patients must have creatinine clearance estimated using the Cockcroft-Gault equation of ≥50 mL/min: Estimated creatinine clearance = (140-age [years]) x weight (kg) (x F)a serum creatinine (mg/dL) x 72, 7) a where F=0.85 for females and F=1 for males, 8) Urine protein: creatinine ratio (UPC) ≤1 OR ≤2+ proteinuria on two consecutive dipsticks taken no less than 1 week apart. Patients with 2+ proteinuria on dipstick must also have UPC <0.5 on 2 consecutive samples. 9) Adequately controlled blood pressure (systolic blood pressure (SBP) ≤140 mmHg; diastolic blood pressure (DBP) ≤ 90mmHg) on maximum of 3 antihypertensive medications. Patients must have a blood pressure (BP) of ≤ 140/90 mmHg taken in the clinic setting by a medical professional within 2 weeks prior to starting study. It is strongly recommended that patients who are on three antihypertensive medications be followed by a cardiologist or a primary care physician for management of BP while on study. 10) Adequately controlled thyroid function, with no symptoms of thyroid dysfunction
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients must have a life expectancy ≥ 16 weeks.
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1. Postmenopausal is defined as: 1) Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments, 2) Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50, 3) radiation-induced oophorectomy with last menses >1 year ago, 4) chemotherapy-induced menopause with >1 year interval since last menses, 5) surgical sterilisation (bilateral oophorectomy or hysterectomy)
* Patients is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
* Patients must have evaluable disease - define as one of the following: 12.1 RECIST 1.1 measurable disease OR, 12.2 Evaluable disease (defined as solid and cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions OR ascites and/or pleural effusion that has been pathologically demonstrated to be disease-related) in the setting of a CA125 > 2 times ULN.
* Formalin fixed, paraffin embedded (FFPE) tumour sample from the primary cancer must be available for central testing. If there is not written confirmation of the availability of an archived tumour sample prior to enrolment the patient is not eligible for the study. For inclusion in i) the optional exploratory genetic research and ii) the optional biomarker research, patients must fulfil the following criteria: 1) Provision of informed consent for genetic research, 2) Provision of informed consent for biomarker research
* If a patient declines to participate in the optional exploratory genetic research or the optional biomarker research, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Previous enrollment or randomization in the present study
* Participation in another clinical study with an investigational product during the last 60 months
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Any previous treatment with poly ADP ribose polymerase(PARP) inhibitor (including olaparib), anti-PD-1, PD-L1, CTLA-4 (including durvalumab and tremelimumab).
* Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma, or other solid tumours including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥5 years. Patients with a history of localised triple negative breast cancer may be eligible, provided they completed their adjuvant chemotherapy more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Resting ECG with Corrected QT Interval(QTc) > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
* Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumour embolization, monoclonal antibodies) ≤21 days prior to the first dose of study drug If sufficient wash-out time has not occurred due to the schedule or Pharmacokinetics(PK) properties of an agent, a longer wash-out period will be required, as agreed by AstraZeneca/MedImmune and the investigator
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug
* Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
* Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria : 1) Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Principal Investigator. 2) Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Principal Investigator.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of Myelodysplastic syndrome/Acute myeloid leukemia(MDS/AML).
* Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female aged 20 years older
Enrollment: 104 (Estimated)
Dates: Start 2018-11-26 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
objective response rate by RECIST 1.1 | 6 months after treatment initiation
  The primary endpoint of the study is objective response rate by RECIST 1.1 (Time frame: up to 6 months after treatment initiation)

SECONDARY OUTCOMES:
Progression-free survival(PFS) | up to 3 years
overall-survival(OS) | up to 3 years
immune-related Response Criteria | up to 3 years
Duration of response | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Yun Lee, MD, Ph.D, Principal Investigator — Severance Hospital
Locations (3):
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol and even raw data will be released after further discussion among researchers.

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Lee JY, Kim BG, Kim JW, Lee JB, Park E, Joung JG, Kim S, Choi CH, Kim HS; Korean Gynecologic Oncology Group (KGOG) investigators. Biomarker-guided targeted therapy in platinum-resistant ovarian cancer (AMBITION; KGOG 3045): a multicentre, open-label, five-arm, uncontrolled, umbrella trial. J Gynecol Oncol. 2022 Jul;33(4):e45. doi: 10.3802/jgo.2022.33.e45. Epub 2022 Mar 4. PMID 35320892
- [Derived] Lee JY, Yi JY, Kim HS, Lim J, Kim S, Nam BH, Kim HS, Kim JW, Choi CH, Kim BG; KGOG investigators. An umbrella study of biomarker-driven targeted therapy in patients with platinum-resistant recurrent ovarian cancer: a Korean Gynecologic Oncology Group study (KGOG 3045), AMBITION. Jpn J Clin Oncol. 2019 Aug 1;49(8):789-792. doi: 10.1093/jjco/hyz085. PMID 31671191